CLINICAL TRIAL: NCT05888909
Title: Multidimensional Accurate Diagnosis and Treatment Technology and Clinical Transformation of Type 2 Diabetes Nephropathy
Status: Recruiting | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Beijing Municipal Science & Technology Commission (Other); China-Japan Friendship Hospital (Other); Beijing Friendship Hospital (Other); Beijing Tongren Hospital (Other); Beijing Hospital (Other Government); Dongzhimen Hospital, Beijing (Other); Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Xiangmei Chen, Professor,Chief physician,Academician of Chinese Academy of Engineering, Chinese PLA General Hospital
Other Study IDs: S2022-482-01
Record Dates: First submitted 2023-05-25; First posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-05

CONDITIONS: Diabetic Nephropathy Type 2; Diabetic Kidney Disease; Type 2 Diabetes
Keywords: Diabetic Nephropathy Type 2; Diabetic Kidney Disease; Type 2 Diabetes; Diagnosis; Treatment
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus, Type 2; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, kidney tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Type 2 diabetic nephropathy: The cohort will be divided into 2 or 3 groups according the pathological results of patients,and at least 3 groups according to clinical features such as renal function and proteinuria.

SUMMARY:
Diabetes nephropathy (DN) is one of the most serious microvascular complications of diabetes, and also an important cause of death and disability of diabetes patients. There is no specific clinical staging of type 2 diabetes nephropathy at home and abroad, and there is no comprehensive study to comprehensively describe the occurrence and development of type 2 diabetes nephropathy through sensitive biomarkers, microvascular disease imaging and functional detection, digital markers and other multi-dimensional diagnosis and evaluation methods. Therefore, our research aims to establish a long-term follow-up queue for the whole cycle of diabetes nephropathy, develop multi-dimensional diagnostic and progress digital markers for diabetes nephropathy, develop a multimodal non-invasive diagnostic model and a new clinical staging/typing, and create a multi-dimensional accurate diagnosis and treatment system for type 2 diabetes nephropathy combining traditional Chinese and western medicine.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years old, regardless of gender; Type 2 diabetes; Having a complete medical history and clinical data; If the patients with type 2 diabetes combined with CKD underwent renal biopsy, the pathological diagnosis should be clear; Patients voluntarily signs an informed consent form.

Exclusion criteria:

Incomplete medical history or clinical data; Patients with hereditary kidney disease; Combined urinary tract infection; Merge autoimmune system diseases; Patients with malignant tumor were expected to survive less than 6 months; Pregnancy and lactation.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Type 2 diabetes and type 2 diabetes patients with CKD
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
change in estimated glomerular filtration rate (eGFR) from baseline | 24months
  eGFR is calculated using the CKD-EPI formula, involving gender, age, and serum creatinine.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, China

REFERENCES:
- [Derived] Wang Q, Dong Z, Zhang W, Zheng Y, Lyu Q, Zhang R, Huang H, Liu F, Wang Y, Zhang L, Cao X, Wu J, Zhou J, Cai G, Chen X. COVID-19 epidemic investigation study of a follow-up cohort of patients with diabetic kidney disease. Front Cell Infect Microbiol. 2024 Aug 20;14:1388260. doi: 10.3389/fcimb.2024.1388260. eCollection 2024. PMID 39228893